CLINICAL TRIAL: NCT02872636
Title: Extracorporeal Filtration of Subarachnoid Hemorrhage Via Spinal Catheter
Acronym: PILLAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minnetronix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DK-0000-001-306
Record Dates: First submitted 2016-08-05; First posted 2016-08-19 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Subarachnoid Hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment Group (Experimental)
  Interventions: Device: Spinal catheter insertion with extracorporeal filtration of CSF

INTERVENTIONS:
Device: Spinal catheter insertion with extracorporeal filtration of CSF — Extracorporeal filtration of CSF

SUMMARY:
The objective of this feasibility study is to demonstrate the safety and feasibility of using an investigational extracorporeal system and catheter to filter hemorrhagic cerebrospinal fluid (CSF) post subarachnoid hemorrhage (SAH) treatment, and reintroduce the CSF via the same catheter.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years or older
* Informed consent by the patient or his/her legally authorized representative
* Modified Fisher Grade 2, 3, or 4
* Hunt & Hess I-III
* First aneurysmal SAH that has been confirmed by Angio, CTA or MRA
* Patient is ≤ 48 hours post bleeding event
* World Federation of Neurosurgeons (WFNS) Grades I-IV and those Grade V patients who improve to Grade IV or less after ventriculostomy.

Exclusion Criteria:

* Patients with a SAH due to mycotic aneurysm or AV malformation
* Patients who present with an acute MI or unstable angina
* Patients with uncontrolled diabetes
* Patients who present with a creatinine > 2.0mg/dl
* Imaging demonstrates supratentorial mass lesions greater than 50 cc
* Imaging demonstrates more than 5 mm of mid-line-shift associated with infarction and or edema
* Effacement of the basilar cisterns (suprasellar, ambient, chiasmatic and quadrageminal)
* Vasospasm on admission as defined by angiographic evidence
* Patients with a coagulopathy that cannot be reversed per the professional discretion of the investigator
* Thrombocytopenia def. platelet count < 100,000
* Patients on low molecular weight heparin e.g., Lovenox
* Patients on Clopidogrel bisulfate (Plavix) or other chronic platelet inhibitors
* Patients with a documented history of cirrhosis
* Patients who will be managed with supportive care rather than intervention
* Obstructive hydrocephalus i.e., non-communicating
* Pregnancy
* History of posterior fusion hardware that would interfere with placement of the catheter
* Pre-existing Lumbar Drain
* Local skin infections or eruptions over the puncture site
* Signs of systemic infection/sepsis or pneumonia
* Lumbar puncture within 6 hours
* Concurrent participation in another study which is not observational or retrospective in nature without prior approval from the Sponsor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-03-23 (Actual); Primary Completion 2018-04-16 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Device/System Safety - Adverse events related to the filtration procedure | 30 days
  Adverse events related to the filtration procedure
Adverse events related to the system catheter insertion | 30 days
  Nerve or tissue damage related to catheter insertion

CONTACTS AND LOCATIONS:
Overall Officials: Julie Messer, Study Director — Minnetronix
Locations (4):
- United States (4):
  - University of Minnesota, Minneapolis, Minnesota
  - Duke University, Durham, North Carolina
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Memorial Hermann, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blackburn SL, Grande AW, Swisher CB, Hauck EF, Jagadeesan B, Provencio JJ. Prospective Trial of Cerebrospinal Fluid Filtration After Aneurysmal Subarachnoid Hemorrhage via Lumbar Catheter (PILLAR). Stroke. 2019 Sep;50(9):2558-2561. doi: 10.1161/STROKEAHA.119.025399. Epub 2019 Jul 26. PMID 31345133